CLINICAL TRIAL: NCT04509362
Title: An 8-Day Initiation Protocol of Advanced Hybrid Closed Loop System In Children and Adolescents With Diabetes Type 1 On Multiple Daily Insulin Injection
Brief Title: An 8-Day Initiation of Advanced Hybrid Closed Loop System In Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Sidra Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 00009930
Record Dates: First submitted 2020-08-01; First posted 2020-08-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Advanced Hybrid Closed Loop System; Minimed 780G; Initiation Protocol
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Advanced Hybrid Closed Loop System — Evaluation of the use of an 8-day structured protocol to initiate patients from MDI to the AHCL system, in achieving safe glycemic control
  Other Names: Minimed 780G

SUMMARY:
One of the available Hybrid closed loop system is MiniMed 670G (Medtronic Diabetes, Northridge, CA, USA), which is indicated for children above 7 years old, adolescents and adults with Type 1 Diabetes. Several studies have shown improved HbA1c, time in target range, and SG variability in children, adolescents and adults with Type 1 Diabetes, where participants were experienced with using CSII therapy, assuming that the success of HCL systems depend on prior use of pump therapy. A recent study, published by diabetes team from Sidra Medicine, Doha has showed that children and adolescents with Type 1 Diabetes on MDI therapy can successfully initiate the HCL system, using a concise structured 10-day protocol, achieving better outcomes than in previous studies, where participants had previous experience with diabetes related technology and longer initiation process.

The AHCL system, Minimed 780G is CE-marked includes additional functionality aiming to provide further protections from highs. The user can choose the algorithm to target a glucose level of 100 or 120 mg/dL. Like for the MiniMed 670G HCL system, users can also choose the algorithm to temporarily target a glucose value of 150 mg/dL. In addition, the AHCL system has the ability to administer correction bolus automatically, targeting 120 mg/dL. The AHCL algorithm was evaluated with a model-based algorithm design platform incorporating a virtual patient simulator, where additional changes were made (lower target ranges and automated correction boluses ( )). A recent study including 12 patients with type 1 diabetes on AHCL system, has shown no episodes of hypoglycemia or diabetic ketoacidosis, while maintaining 99% time spent in closed loop and high time in ra1]\nge ( ). AHCL decreased Auto Mode exits and alerts, and improves glycaemia without compromising safety, despite multiple food and exercise challenges ( ).

Sidra Medicine is the only center for childhood diabetes in Qatar. Around 80% of type 1 diabetes patients are using a device (insulin pump/glucose sensor) and around 45% are using sensor-augmented pump (SAP)/HCL systems.

DETAILED DESCRIPTION:
This study is a single-arm, single-center, clinical investigation in subjects with type 1 diabetes on AHCL insulin pump in a period of 3 months.

The study will include an 9-month extension phase, to which participants may voluntarily decide to take part in, cumulating a total of one-year period duration. Visits wil be scheduled every 3 months, as per routine practice. TIR, HbA1c, demographics and clinical data will be analyzed on 3 months period.

A total of 33 subjects (age 7-17 years) will be enrolled in order to reach 30 subjects who will complete the 3 months study.

After reviewing the patient's eligibility and interest, the investigators will obtain informed consent and assent as appropriate. The investigators will start the clinical process for initiating an insulin pump, which is typically done with pre-pump classes. A clinically obtained HbA1c assessment will be performed via fingerstick and DCA 2000 at baseline and 3 months during the study.

Collection of demographics and medical history, data for diabetes devices (eg meters, sensors, pumps) and brief clinical physical exam including vital signs and skin assessment will be obtained via Hospital Electronic Medical File (Cerner Millennium) and will be kept as electronic data on a separate research server.

The different continuous baseline values will be checked for normality of distribution using the mean-median comparison, skewness and kurtosis (-3 to +3), spread, Kolmogorov-Smirnow and Shapiro-Wild tests, outliers, histograms and Q-Q-plots.

The initiation protocol consisted of four main stages: AHCL system compatibility assessment, AHCL system training, Manual Mode and Auto Mode stages.

Step 1. AHCL system compatibility assessment

Step 1 will be used to select participants for the study, based on inclusion and exclusion criteria (explained below) as well as patients' interest. It consists of 2 sessions:

AHCL System Introduction session (Clinic visit), one-hour duration (groups of 8-12 patients), where the AHCL system will be explained. Individuals' responsibilities (e.g. bolusing before meal, calibrating the system 3-4 times per day, responding to alerts and alarms, downloading pump data from home) and expectations (e.g. improvements in glycemic control, less glucose variability, hypoglycemia minimization, workload of diabetes management) will be discussed.

AHCL System readiness session, 1-hour duration, where evaluation will be performed on carb counting, bolus for carbs and correction, SMBG. Participants will send food log diary and phone call consultation will be performed.

Step 2: AHCL system training

A similar approach currently used in Sidra for MiniMed 670G system initiation will be used in the study. AHCL system training will be performed in groups (three to five individuals and their parents/guardians). The program includes three sessions of two to three hours on three consecutive days. CGM will be initiated the first day of the training, for education and observational purposes and for baseline data collection (no insulin delivery by the pump) Details are explained in the table:

Each session will be provided by two educators from 12pm to 3pm. Timing of the long acting insulin injection will be moved two hours ahead each day during training sessions, to reach 12pm the day before the HCL system initiation in Manual Mode, to avoid the use of temporary basal at insulin pump initiation.

Step 3: Manual Mode Participants will initiate the use of the AHCL system in Manual Mode (Clinic visit) with suspend before low feature for 72 hours to allow the algorithm to collect insulin utilization and CGM data to establish personalized Auto Mode initiation parameters. Sidra's validated protocol for SAP initiation (Auto-Generator app), also used in 10-day initiation protocol, with review of CGM data (step 2) will be used: in short, the protocol inputs the current insulin program (MDI), calculates a 10 to 20% reduction of total daily dose, with a 40/60 basal/bolus distribution in four or five basal rates. Insulin to carbohydrate ratio (ICR) settings utilizes the formula of 300-450/Total Daily dose (TDD) and, the formula of 90-110/TDD (mmol/l) with two CF settings, the nighttime CF factor is set 10-20% higher than the daytime CF. Active insulin is set time (3 hours), suspend before low feature is turned on with a threshold of 3.0-3.8 mmol/l (55-70 mg/dl) and glucose target range from 5.0 mmol/l to 7.2 mmol/l (90-130 mg/dl).

Step 4: Auto Mode The Auto Mode feature of the AHCL system will be activated 72 hours after manual mode initiation (virtual visit, using Skype Meet) and will be used continuously for 84 days.

The patient/family will upload data into the CareLink system, and the data will be reviewed by a member of the clinical team. Adjustments to system settings will be suggested to the family as clinically appropriate. The rationale for system setting adjustments will be documented.

Follow up visits will be performed on 7, 14, 28 days of aHCL initiation. After the first month of aHCL system, visits will be every three months during the study.

HbA1c will be obtained using point of care DCA Vantage Analyzer (Siemens, Erlangen, Germany) at baseline and at the end of the study.

The study will submit the proposal to Local and National Ethics Committee in Qatar to get Ethical approval before commencing the study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes >1 year prior to consent date. Diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. HbA1c < 12.5%
3. Age 7-17 years at the initiation of the system
4. Multiple Daily Injections (Basal Bolus therapy) with Total daily insulin use of great than 8.0 units per day over a 1-week period
5. Willing and able (access to internet from home) to download information into the Medtronic CareLink software
6. Clinically able to start the AHCL system
7. History of 3 clinic visits in the last year

Exclusion Criteria:

1. DKA in the 6 months prior to screening visit
2. Pregnancy
3. Untreated diabetes retinopathy, or other causes that ,in the investigator's opinion, precludes the individual from participating in the trial.

Ages: 7 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants with Type 1 Diabetes, on multiple daily injections, using self-monitoring of blood glucose or continuous glucose monitoring, no prior pump experience.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
TIR (70-180 mg/dl) | 3 months
  Change from baseline to the first 3 months
TIR (70-180 mg/dl | 12 months
  Change from baseline to the 12 months

SECONDARY OUTCOMES:
HbA1c change | 3 months
  Change in HbA1c from Baseline to 3 months
HbA1c change | 12 months
  Change in HbA1c from Baseline to 12 months
Sensor glucose wear | 3 months
  Change in Sensor glucose wear from Baseline to 3 months
Sensor glucose wear | 12 months
  Change in Sensor glucose wear from Baseline to 12 months
Auto Mode Usage | 3 months
  Change in Auto Mode Usage from Baseline to 3 months
Auto Mode Usage | 12 months
  Change in Auto Mode Usage from Baseline to 12 months
Severe Hypoglycemia | 3 months
  Number of events in the first 3 months
Severe Hypoglycemia | 12 months
  Number of events in the 12 months
Diabetic Ketoacidosis | 3 months
  Number of events in the first 3 months
Diabetic Ketoacidosis | 12 months
  Number of events in 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sidra Medicine, Doha, Qa, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
It depends on Institution decision, waiting response

REFERENCES:
- [Background] Garg SK, Weinzimer SA, Tamborlane WV, Buckingham BA, Bode BW, Bailey TS, Brazg RL, Ilany J, Slover RH, Anderson SM, Bergenstal RM, Grosman B, Roy A, Cordero TL, Shin J, Lee SW, Kaufman FR. Glucose Outcomes with the In-Home Use of a Hybrid Closed-Loop Insulin Delivery System in Adolescents and Adults with Type 1 Diabetes. Diabetes Technol Ther. 2017 Mar;19(3):155-163. doi: 10.1089/dia.2016.0421. Epub 2017 Jan 30. PMID 28134564
- [Background] Grosman B, Wu D, Miller D, Lintereur L, Roy A, Parikh N, Kaufman FR. Sensor-Augmented Pump-Based Customized Mathematical Model for Type 1 Diabetes. Diabetes Technol Ther. 2018 Mar;20(3):207-221. doi: 10.1089/dia.2017.0333. PMID 29565722
- [Background] Paldus B, Lee MH, Jones HM, McAuley SA, Horsburgh JC, Roem KL, Ward GM, MacIsaac RJ, Cohen N, Colman PG, Jenkins AJ, O'Neal DN. Glucose Control Using a Standard Versus an Enhanced Hybrid Closed Loop System: A Randomized Crossover Study. Diabetes Technol Ther. 2019 Jan;21(1):56-58. doi: 10.1089/dia.2018.0279. PMID 30620641
- [Result] Thabit H, Hovorka R. Coming of age: the artificial pancreas for type 1 diabetes. Diabetologia. 2016 Sep;59(9):1795-805. doi: 10.1007/s00125-016-4022-4. Epub 2016 Jun 30. PMID 27364997
- [Result] Biester T, Nir J, Remus K, Farfel A, Muller I, Biester S, Atlas E, Dovc K, Bratina N, Kordonouri O, Battelino T, Philip M, Danne T, Nimri R. DREAM5: An open-label, randomized, cross-over study to evaluate the safety and efficacy of day and night closed-loop control by comparing the MD-Logic automated insulin delivery system to sensor augmented pump therapy in patients with type 1 diabetes at home. Diabetes Obes Metab. 2019 Apr;21(4):822-828. doi: 10.1111/dom.13585. Epub 2018 Dec 21. PMID 30478937
- [Result] U.S. Food and Drug Administration (2019) FDA approves first automated insulin delivery device for type 1 diabetes. Available from www.fda.gov/news-events/press-announcements/fda-approves-first-automated-insulin-delivery-device-type-1-diabetes. Accessed 21 March 2019
- [Result] Weaver KW, Hirsch IB. The Hybrid Closed-Loop System: Evolution and Practical Applications. Diabetes Technol Ther. 2018 Jun;20(S2):S216-S223. doi: 10.1089/dia.2018.0091. Epub 2018 Jun 6. PMID 29873517
- [Result] Trevitt S, Simpson S, Wood A. Artificial Pancreas Device Systems for the Closed-Loop Control of Type 1 Diabetes: What Systems Are in Development? J Diabetes Sci Technol. 2016 May 3;10(3):714-23. doi: 10.1177/1932296815617968. Print 2016 May. PMID 26589628
- [Result] Forlenza GP, Pinhas-Hamiel O, Liljenquist DR, Shulman DI, Bailey TS, Bode BW, Wood MA, Buckingham BA, Kaiserman KB, Shin J, Huang S, Lee SW, Kaufman FR. Safety Evaluation of the MiniMed 670G System in Children 7-13 Years of Age with Type 1 Diabetes. Diabetes Technol Ther. 2019 Jan;21(1):11-19. doi: 10.1089/dia.2018.0264. Epub 2018 Dec 26. PMID 30585770
- [Result] Petrovski G, Al Khalaf F, Campbell J, Fisher H, Umer F, Hussain K. 10-Day structured initiation protocol from multiple daily injection to hybrid closed-loop system in children and adolescents with type 1 diabetes. Acta Diabetol. 2020 Jun;57(6):681-687. doi: 10.1007/s00592-019-01472-w. Epub 2020 Jan 17. PMID 31953687